CLINICAL TRIAL: NCT07219654
Title: A Phase 2, Double-blinded, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Allogeneic Dermal Fibroblasts (TPX-115) in Patients With Partial-thickness Rotator Cuff Tear
Brief Title: Efficacy and Safety Study of TPX-115 on Partial-thickness Rotator Cuff Tear
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tego Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TG-TPX-115-24-US-01
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Partial Thickness Rotator Cuff Tears
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- TPX-115 low dose (Experimental)
  Interventions: Biological: TPX-115
- TPX-115 medium dose (Experimental)
  Interventions: Biological: TPX-115
- TPX-115 high dose (Experimental)
  Interventions: Biological: TPX-115
- Cryopreserving hyaluronic acid medium (Experimental)
  Interventions: Other: Cryopreserving hyaluronic acid medium
- saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: TPX-115 — Single injection of Allogeneic dermal fibroblasts (TPX-115) via ultrasound-guided intratendinous injection
  Arms: TPX-115 high dose; TPX-115 low dose; TPX-115 medium dose
Other: Cryopreserving hyaluronic acid medium — Medium included in TPX-115 for cryopreservation
  Arms: Cryopreserving hyaluronic acid medium
Drug: Saline — Saline
  Arms: saline

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of allogeneic dermal fibroblasts (TPX-115) compared to placebo in patients with Partial-Thickness Rotator Cuff Tear(PTRCT).

Primary endpoint is to evaluate the efficacy of TPX-115 compared to placebo, as measured by improvement in the Constant-Murley Score (CMS) in patients with PTRCT.

Secondary endpoints are:

* To evaluate functional (including shoulder pain) and structural improvements in the affected shoulder after administration of TPX-115 compared to placebo in patients with PTRCT
* To evaluate the safety and tolerability of TPX-115 in patients with PTRCT
* To assess the immunogenicity of TPX-115

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >= 18 years.
* Patients with PTRCT involving <= 50% of the tendon thickness based on depth of defect (or Grade I or II on Ellman classification) assessed by MRI within the last 3 months prior to screening and determined by the investigator.
* Patients with clinical symptoms including but not limited to pain, muscle weakness, or limited active range of motion (ROM) of PTRCT persisting for more than 3 months despite conservation treatment.
* Patients who report a usual pain level of >= 4 on visual analogue scale (VAS) at screening.
* Patients who had, in the opinion of the investigator, at least 1 reasonable physical therapy course and no substantial response within 6 months prior to enrollment.
* Patients who are willing to discontinue all pain medications on the shoulder (except rescue medication of < 3.25g acetaminophen per day) at least 72 hours prior to screening and throughout the duration of study.
* Patients in general good health, with no concomitant conditions or taking treatments potentially representing confounding factors and interfering with the study treatment or study procedures and their results or putting the patient at a greater risk, as per the investigator's documented clinical judgment.
* Patients who meet the following laboratory criteria, with results within 5% of the specified normal reference ranges:

  1. Hemoglobin: 12 to 18 g/dL.
  2. White Blood Cell (WBC) Count: 4.5 to 11.0 x 10^3/uL.
* Patients with eGFR > 60 ml/min
* Patients with ALT and AST < 3xUpper limit of normal
* Patients who are willing and able to give written informed consent for participation in the study.

Exclusion Criteria:

* Patients with full-thickness rotator cuff tear in the affected shoulder as assessed by MRI.
* Patients with both partial- and full-thickness rotator cuff tear in the affected shoulder.
* Patients who have experienced previous surgeries in the affected shoulder within 12 months prior to enrollment.
* Patients who have received subacromial or intra-articular injection in the affected shoulder within 3 months prior to screening visit.
* Patients who have a history of cell therapy or prolotherapy in the affected shoulder.
* Patients who have received platelet-rich plasma (PRP) injection in the affected shoulder within 6 months prior to screening visit.
* Patients who have received systemic immunosuppressive therapy within 4 weeks prior to screening visit.
* Patients who have any of the following clinically significant diseases at screening or have medical history of past:

  1. inflammatory joint disease (eg, septic arthritis, rheumatoid inflammation)
  2. other shoulder disease, in the affected shoulder, that may cause shoulder pain or functional disorder (eg, arthritis, cervical spine disorders, subacromial pathological morphology leading to impingement syndrome)
  3. autoimmune disease
  4. active hepatitis B or C (except for simple carriers and hepatitis B patients with antiviral medications for 6 months before screening)
  5. human immunodeficiency virus antibody-positive
  6. history of systemic malignancy within the last 5 years
  7. coagulopathy
  8. genetic disorders affecting fibroblasts or collagen production (eg. achondroplasia, osteogenesis imperfecta)
  9. other serious diseases (eg. neurological cardiovascular, renal or hepatic disease, uncontrolled diabetes, etc) that, inthe opinion of the investigator, might confound study results or pose additional risk to the patient by their participation in the study.
* Female patients who are pregnant or breastfeeding.
* Female patients planning pregnancy during the study period. Women of childbearing potential who do not agree to maintain contraception, or who do not agree to use the appropriate method of contraception (ie, double effective barrier contraception) during the study period.

Note: Suitable contraceptive methods are condom, sponge, gel, diaphragm for contraception, hormonal contraceptives, intrauterine device, etc. Periodic abstinence (eg, calendar method, ovulation method, symptom body temperature method, post-ovulation method) and restraint are not considered an accepted method of contraception. However, women unable to become pregnant due to menopause (at least 12 months since last menstrual period) can participate in the study with negative pregnancy test results.

* Patients who have administered other IPs or devices within 4 weeks or 5 half-lives, whichever is greater, prior to the IP administration.
* Patients whom the principal investigator considers inappropriate for the study due to any other reasons than those listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Constant-Murley Score(CMS) at Week 24 | Baseline, Week 24
  The CMS is calculated from 0 (worst function) to 100 (best function) points

SECONDARY OUTCOMES:
Change from baseline in Constant-Murley Score(CMS) at Weeks 4, 12, and 52 | Baseline, Week 4, Week 12, Week 52
  The CMS is calculated from 0 (worst function) to 100 (best function) points
Increase of at least 8 points from baseline in Constant-Murley Score(CMS) at Week 24 | Baseline, Week 24
  The CMS is calculated from 0 (worst function) to 100 (best function) points
Change from baseline in Visual Analogue Scale(VAS) (0 to 10 cm) score for shoulder pain at Weeks 4, 12, 24, and 52 | Baseline, Week 4, Week 12, Week 24, Week 52
  The VAS is a horizontal line, 10 cm in length, with anchor statements on the left (0 cm; meaning 'no pain') and on the right (10cm; meaning 'extreme pain')
Change from baseline in Range of Motion(ROM) in the affected shoulder at Weeks 4, 12, 24, and 52 | Baseline, Week 4, Week 12, Week 24, Week 52
Change from baseline in American Shoulder and Elbow Surgeons(ASES) score at Weeks 4, 12, 24, and 52 | Baseline, Week 4, Week 12, Week 24, Week 52
  The ASES score is calculated from zero (worst) to 100 (best) points
Change from baseline in Simple Shoulder Test at Weeks 4, 12, 24, and 52 | Baseline, Week 4, Week 12, Week 24, Week 52
Change from baseline in tear size (mm) on MRI at Week 52 | Baseline, Week 52
Change from baseline in tendon thickness (mm) on MRI at Week 52 | Baseline, Week 52
Change from baseline in tear/footprint (%p) on MRI at Week 52 | Baseline, Week 52
Change from baseline in tendinosis on MRI at Week 52 | Baseline, Week 52
  The grade of tendinosis is assessed from zero (normal) to 3 (marked) by a central reader only (independent evaluator).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - BioSolutions Clinical Research Center, La Mesa, California
  - Sports & Orthopedic Center - Advanced Research, Deerfield Beach, Florida
  - Rush University Medical Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Undecided